CLINICAL TRIAL: NCT04310709
Title: Phase II Study of Regorafenib-nivolumab Combination Therapy for Chemotherapy-naïve Patients With Unresectable or Metastatic Hepatocellular Carcinoma
Brief Title: Combination of Regorafenib and Nivolumab in Unresectable Hepatocellular Carcinoma
Acronym: RENOBATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, Changhoon Yoo, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RENOBATE
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Carcinoma, Hepatocellular; Hepatoma
Keywords: Hepatocellular carcinoma; Regorafenib; Nivolumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REGONIVO (Experimental): Nivolumab - 480 mg IV on Day 1, every 4 weeks
  Regorafenib
  - 80 mg per oral once daily for 21 consecutive days starting on Day 1, every 4 weeks.
  Interventions: Drug: Regorafenib/Nivolumab

INTERVENTIONS:
Drug: Regorafenib/Nivolumab — Combination of regorafenib and nivolumab

SUMMARY:
Regorafenib and nivolumab are proven effective agents for the management of unresectable hepatocellular carcinoma patients. As preclinical studies have suggested potential synergism between antiangiogenic agents and immune checkpoint inhibitors, regorafenib and nivolumab may have synergism in terms of efficacy. Herein, this study investigates the combination of regorafenib and nivolumab as first-line therapy in patients with unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years at time of signing Informed Consent Form
2. Ability to comply with the study protocol, in the investigator's judgment
3. HCC that was histologically/cytologically confirmed or clinically diagnosed by AASLD criteria in cirrhotic patients. Patients without liver cirrhosis require histological confirmation of HCC
4. Locally advanced unresectable or metastatic disease that is not amenable to curative surgical and/or locoregional therapies, or that progressed after surgical and/or locoregional therapies
5. No prior systemic therapy for HCC
6. At least one measurable (per RECIST 1.1) lesion as confirmed by imaging within 28 days prior to initiation of study treatment
7. Patients who received prior local therapy (e.g., radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, transarterial chemoembolization, transarterial embolization, etc.) are eligible provided that other target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST 1.1.
8. Pre-treatment tumor tissue sample (if available)

   * If tumor tissue is available, approximately 10 to 30 slides containing unstained, freshly cut, serial sections will be required subsequently for translational research.
   * If tumor tissue is not available (e.g., depleted because of prior diagnostic testing), patients are still eligible.
9. ECOG Performance Status score 0 or 1
10. Child-Pugh class A
11. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment, unless otherwise specified:

    * ANC ≥ 1.0 x 109/L (1000/microL) without granulocyte colony-stimulating factor support
    * Platelet count ≥ 75 x 109/L (75,000/mciroL) without transfusion
    * Hemoglobin ≥ 90 g/L (9 g/dL): Patients may be transfused to meet this criterion.
    * AST, ALT, and alkaline phosphatase (ALP) ≥ 3 x upper limit of normal (ULN)
    * Serum bilirubin ≥ 2 x ULN
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula)
    * Serum albumin ≥ 28 g/L (2.8 g/dL)
    * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 2 x ULN
    * Urine dipstick for proteinuria < 2+
    * Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours.
12. Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to Grade ≤ 1 prior to study entry, with the exception of alopecia
13. Negative HIV result at screening test or prior tested conducted within 3 years
14. Documented virology status of hepatitis, as confirmed by screening HBV and HCV serology test

    - Patients with active hepatitis B virus (HBV) must meet the followings: HBV DNA < 500 IU/mL obtained within 14 days prior to initiation of study treatment, anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study
15. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons)#1 must agree to use contraception#2 from the time of informed consent until 5 months or more after the last dose of the investigational product. Also, women must agree not to breastfeed from the time of informed consent until 5 months or more after the last dose of the investigational product.
16. Men must agree to use contraception #2 from the start of study treatment until 7 months or more after the last dose of the investigational product.

Exclusion Criteria:

1. Patients who are diagnosed with fibrolamellar HCC, sarcomatoid HCC, or combined type of cholangiocarcinoma and HCC
2. Patients with a history of malignancy other than HCC within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, and Stage I uterine cancer
3. Patients with a history of leptomeningeal seeding
4. Patients with symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

   * Asymptomatic patients with treated CNS lesions are eligible, provided that all of the following criteria are met:

     1. The patients must have at least one measurable lesion, per RECIST 1.1, other than CNS metastases
     2. The patient must not have a history of intracranial hemorrhage or spinal cord hemorrhage
     3. The metastatic lesions have to be limited in cerebellum or supratentorial region (e.g., not to the midbrain, pons, medulla, or spinal cord)
     4. There must be no evidence of interim progression between the completion of CNS-directed therapy and initiation of the study treatment
     5. The patient must not undergo stereotactic radiotherapy within 7 days, whole-brain radiotherapy within 14 days, or neurosurgical resection within 28 days prior to initiation of the study treatment
     6. The patient must not have ongoing requirement for corticosteroids for CNS disease
   * Anticonvulsant therapy at a stable dose is permitted.
   * Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan.
5. Patients with current of past history of autoimmune disease or immunodeficient disease (including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis) with the following exceptions:

   * Patients with autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible.
   * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible.
   * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

     1. Rash must cover < 10% of body surface area
     2. Disease has to be well controlled at baseline and requires only low-potency topical corticosteroids
     3. There must be no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
6. Patients with current or past history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

   - Patients with history of radiation pneumonitis in the radiation field (fibrosis) are eligible if the radiation pneumonitis has been confirmed as stable (beyond acute phase) without any concerns about recurrence.
7. Patients who have experienced a transient ischemic attack, cerebrovascular accident, thrombosis, or thromboembolism (pulmonary arterial embolism or deep vein thrombosis) within 6 months before initiation of study treatment
8. Patients with a history of uncontrollable or significant cardiovascular disease meeting any of the following criteria:

   * Myocardial infarction within 6 months before initiation of study treatment
   * Uncontrollable angina pectoris within 6 months before initiation of study treatment
   * New York Heart Association Class II or greater congestive heart failure within 6 months before initiation of study treatment
   * Uncontrollable hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150 mmHg or diastolic blood pressure > 90 mmHg based on an average of ≥ 3 BP readings on ≥ 2 sessions)
   * Arrhythmia requiring treatment
9. Patients with congenital long QT syndrome or corrected QT interval >450 ms (calculated with use of the Fridericia method) at screening
10. Patients with systemic infections (including active tuberculosis) requiring treatment
11. Patients with history of hypertensive crisis or hypertensive encephalopathy
12. Patients with significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of study treatment
13. Patients who underwent major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment or who are expected to need a major surgical procedure during the study
14. Patients who have received radiotherapy within 28 days before initiation, or radiotherapy to bone metastases within 14 days before initiation
15. Patients with prior history of allogeneic stem cell or solid organ transplantation
16. Patients with current or past history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
17. Patients with untreated or incompletely treated varices with active bleeding or high risk for bleeding
18. Patients with moderate or severe ascites
19. Patients with history of hepatic encephalopathy
20. Patients with evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
21. Patients who had recent (within 10 days of first dose of study treatment) use of aspirin (> 300 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol
22. Patients who had recent use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose

    * Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR < 1.5 x ULN and aPTT within normal limits within 14 days prior to initiation of study treatment.
    * Prophylactic use of low molecular-weight heparin (i.e., enoxaparin 40 mg/day) is allowed.
23. Patients who treated with strong CYP3A4 inducers within 14 days prior to initiation of study treatment, including rifampin (and its analogues) or St. John's wort
24. Patients who have previously received CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
25. Patients who were treated with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
26. Patients who were treated with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received temporary, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
    * Patients who received mineralocorticoids (e.g., fludrocortisone), or corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
27. Patients who had abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to initiation of study treatment
28. Patients who had intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding within 6 months prior to initiation of study treatment

    - Patients with signs/symptoms of sub-/occlusive syndrome/intestinal obstruction at time of initial diagnosis may be enrolled if they had received definitive (surgical) treatment for symptom resolution.
29. Women who are pregnant or breastfeeding, or possibly pregnant
30. Other patients judged by the investigator or sub-investigator to be inappropriate as subjects of this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months
  Proportion of patients with complete response/partial response graded by Response Criteria in Solid Tumor version 1.1

SECONDARY OUTCOMES:
Adverse events | 1 year
  Proportion of patients experiencing adverse events graded by National Cancer Institute Common Terminology Criteria version 5.0
Progression-free survival | 1 year
  Time between the start of study treatment and progressive disease or any cause of death
Overall survival | 1 year
  Time between the start of study treatment and any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, MD, PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Bundang CHA Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruix J, Qin S, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Breder V, Gerolami R, Masi G, Ross PJ, Song T, Bronowicki JP, Ollivier-Hourmand I, Kudo M, Cheng AL, Llovet JM, Finn RS, LeBerre MA, Baumhauer A, Meinhardt G, Han G; RESORCE Investigators. Regorafenib for patients with hepatocellular carcinoma who progressed on sorafenib treatment (RESORCE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Jan 7;389(10064):56-66. doi: 10.1016/S0140-6736(16)32453-9. Epub 2016 Dec 6. PMID 27932229
- [Background] Yoo C, Park JW, Kim YJ, Kim DY, Yu SJ, Lim TS, Lee SJ, Ryoo BY, Lim HY. Multicenter retrospective analysis of the safety and efficacy of regorafenib after progression on sorafenib in Korean patients with hepatocellular carcinoma. Invest New Drugs. 2019 Jun;37(3):567-572. doi: 10.1007/s10637-018-0707-5. Epub 2018 Dec 7. PMID 30523474
- [Background] Yoo C, Ryu YM, Kim SY, Kim J, Ock CY, Ryu MH, Kang YK. Association between the exposure to anti-angiogenic agents and tumour immune microenvironment in advanced gastrointestinal stromal tumours. Br J Cancer. 2019 Nov;121(10):819-826. doi: 10.1038/s41416-019-0596-1. Epub 2019 Oct 14. PMID 31607749
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Derived] Kim HD, Jung S, Lim HY, Ryoo BY, Ryu MH, Chuah S, Chon HJ, Kang B, Hong JY, Lee HC, Moon DB, Kim KH, Kim TW, Tai D, Chew V, Lee JS, Finn RS, Koh JY, Yoo C. Regorafenib plus nivolumab in unresectable hepatocellular carcinoma: the phase 2 RENOBATE trial. Nat Med. 2024 Mar;30(3):699-707. doi: 10.1038/s41591-024-02824-y. Epub 2024 Feb 19. PMID 38374347